CLINICAL TRIAL: NCT00000517
Title: Boston Area Anticoagulation Trial for Atrial Fibrillation (BAATAF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, J. Philip Kistler, Physician, Massachusetts General Hospital
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 36; R01HL033233-06 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Arrhythmia; Atrial Fibrillation; Cardiovascular Diseases; Cerebral Embolism and Thrombosis; Cerebrovascular Disorders; Heart Diseases; Thrombophlebitis; Cerebrovascular Accident
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Cardiovascular Diseases; Intracranial Embolism and Thrombosis; Cerebrovascular Disorders; Heart Diseases; Thrombophlebitis; Stroke | interventions — Warfarin

INTERVENTIONS:
Drug: warfarin

SUMMARY:
To determine the benefits and risks of oral anticoagulant therapy in reducing embolic stroke and systemic emboli in patients with atrial fibrillation without rheumatic heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

The efficacy of oral anticoagulation therapy in reducing the risk of embolic stroke in patients with atrial fibrillation and rheumatic heart disease was well known. The value of anticoagulant therapy in patients with atrial fibrillation without rheumatic heart disease had not been established. Several studies strongly suggested that although the risk of stroke in patients with atrial fibrillation was greatest in the presence of valvular disease, the risk of stroke in the absence of valvular disease was also much greater in patients with atrial fibrillation than those without this arrhythmia. What was lacking was a detailed controlled study assessing the degree of reduction in stroke risk by anticoagulation of fibrillating patients without valvular disease.

The second question asked was whether the added potential morbidity or mortality associated with long-term anticoagulation therapy justified its use in the prophylactic treatment of neurologically asymptomatic patients with atrial fibrillation, even if it did reduce stroke risk. Gastrointestinal, urinary tract, cutaneous and joint hemorrhages were all potential serious complications, as was cerebral hemorrhage, including bleeding into areas of recent cerebral infarction. Interest had again focused on hemorrhagic complications of stroke in anticoagulated patients and among risk factors for hemorrhage were large, recent infarcts. No one suggested that anticoagulation, even if very successful in reducing stroke risk, would eliminate it altogether, and thus hemorrhagic infarction was an important potential problem, as was assessment of risk of primary intracerebral hemorrhage.

DESIGN NARRATIVE:

Randomized non-blind. Recruitment began in September 1985 and ended in June 1989. The experimental group of 212 patients received long-term, low-dose warfarin. The control group of 208 patients did not receive warfarin but could choose to take aspirin. Average follow-up was 2.2 years. The primary endpoint was non-hemorrhage stroke. At entry and annually, the history was recorded and patients underwent a physical examination focusing on neurologic factors. Every year, beginning at six months, patients were sent a questionnaire on neurologic symptoms, bleeding episodes, and other medical conditions. Study nurses contacted all patients to review their responses. Each patient's referring physician was contacted at three months and nine months during each year of follow-up.

Participating institutions in the multicenter trial were organized into three groups. At Group I institutions, on-site investigators performed all clinical evaluations. In Group II, personnel from the central site hospital, the Massachusetts General Hospital, traveled to the local hospitals to evaluate, randomize, and follow patients. Group III institutions referred patients directly to the Massachusetts General Hospital for all procedures.

ELIGIBILITY:
Men and women, 18 years of age or older, with non-rheumatic atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1985-07; Primary Completion 1991-06 (Actual); Study Completion 1991-06 (Actual)

REFERENCES:
- [Background] Boston Area Anticoagulation Trial for Atrial Fibrillation Investigators; Singer DE, Hughes RA, Gress DR, Sheehan MA, Oertel LB, Maraventano SW, Blewett DR, Rosner B, Kistler JP. The effect of low-dose warfarin on the risk of stroke in patients with nonrheumatic atrial fibrillation. N Engl J Med. 1990 Nov 29;323(22):1505-11. doi: 10.1056/NEJM199011293232201. PMID 2233931
- [Background] Lancaster TR, Singer DE, Sheehan MA, Oertel LB, Maraventano SW, Hughes RA, Kistler JP. The impact of long-term warfarin therapy on quality of life. Evidence from a randomized trial. Boston Area Anticoagulation Trial for Atrial Fibrillation Investigators. Arch Intern Med. 1991 Oct;151(10):1944-9. PMID 1929681
- [Background] Singer DE, Hughes RA, Gress DR, Sheehan MA, Oertel LB, Maraventano SW, Blewett DR, Rosner B, Kistler JP. The effect of aspirin on the risk of stroke in patients with nonrheumatic atrial fibrillation: The BAATAF Study. Am Heart J. 1992 Dec;124(6):1567-73. doi: 10.1016/0002-8703(92)90074-6. PMID 1462916
- [Background] Kistler JP, Singer DE, Millenson MM, Bauer KA, Gress DR, Barzegar S, Hughes RA, Sheehan MA, Maraventano SW, Oertel LB, et al. Effect of low-intensity warfarin anticoagulation on level of activity of the hemostatic system in patients with atrial fibrillation. BAATAF Investigators. Stroke. 1993 Sep;24(9):1360-5. doi: 10.1161/01.str.24.9.1360. PMID 8362431